CLINICAL TRIAL: NCT06934733
Title: The Efficacy of Oral Cryotherapy in Preventing TROP2-ADC-Induced Oral Mucositis in Patients With Advanced Breast Cancer: A Randomized, Controlled, Multicenter Clinical Study
Brief Title: The Efficacy of Oral Cryotherapy in Preventing TROP2-ADC-Induced Oral Mucositis in Patients With Advanced Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HNCH-MBC17
Record Dates: First submitted 2025-03-27; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral cryotherapy (Experimental)
  Interventions: Other: Oral cryotherapy
- Routine oral care (Other)
  Interventions: Other: Routine oral care

INTERVENTIONS:
Other: Oral cryotherapy — Patients randomly assigned to the experimental group underwent TROP2-ADC treatment. They continuously held ice cubes and ice water from 15 minutes before the infusion, throughout the infusion process, and for 15 minutes after the infusion. Ice cubes were promptly replaced with fresh ones as they melted. Patients were instructed not to consume any food or liquids orally for 1 hour following the completion of the ice therapy.
  Arms: Oral cryotherapy
Other: Routine oral care — Patients in the control group did not receive oral cryotherapy during the TROP2-ADC infusion but only received routine oral care.
  Arms: Routine oral care

SUMMARY:
The incidence of oral mucositis associated with TROP2-ADC therapy in patients with advanced breast cancer is notably high. Identifying effective preventive and therapeutic strategies is essential for enhancing patient quality of life and optimizing treatment outcomes. Oral cryotherapy has been demonstrated to be efficacious in mitigating oral mucositis induced by radiotherapy and chemotherapy. Consequently, this study seeks to investigate the potential preventive efficacy of oral cryotherapy on TROP2-ADC-induced oral mucositis in patients with advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily enrolled in the study, signed the informed consent form, and demonstrated good compliance.
2. Age ≥ 18 years at the time of informed consent signing.
3. Patients with locally advanced or recurrent/metastatic breast cancer receiving TROP2-ADC treatment for the first time.
4. ECOG PS: 0-2 points;
5. The expected survival time was more than 3 months;
6. Adequate organ and bone marrow function, with no transfusions or treatments with recombinant human thrombopoietin or colony-stimulating factors within 1 week before the first dose, is defined as follows:

   1. Blood routine: Neutrophil count (NEUT#) ≥ 1.5×109/L; Platelet (PLT) ≥ 75×109/L; Hemoglobin ≥ 90g/L
   2. Liver function: AST and ALT ≤ 3 × ULN; for patients with liver metastasis, AST and ALT ≤ 5 × ULN.
   3. Renal function: Creatinine ≤ 1.5 × ULN or Ccr ≥ 60 ml/min (Cockcroft-Gault formula provided).
   4. Cardiac function: LVEF ≥ 50% by ECHO or MUGA scan.
7. Patients with a negative pregnancy test and reproductive potential must agree to use effective non-hormonal contraception during treatment and for at least 3 months after the last dose of the investigational drug.
8. Voluntary participants who sign informed consent, demonstrate good compliance, and agree to follow-up.

Exclusion Criteria:

1. Prior TROP2-targeted treatment was administered.
2. Patients with active oral mucositis or oral ulcers were excluded.
3. Patients with serious concomitant diseases, as judged by researchers, that threaten safety or impede study completion, including uncontrolled hypertension, severe diabetes, and active infections, were excluded.
4. Other conditions where the investigator determines the patient is unsuitable for study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of oral mucositis within 8 weeks (scored according to the CECAE 5.0 standard) | From the start of TROP2-ADC treatment to the 8th week
  The incidence and severity of oral mucositis at week 8

SECONDARY OUTCOMES:
The incidence and severity of oral mucositis at week 12 and week 24 | From the start of TROP2-ADC treatment to the 12th and 24th week
  The incidence and severity of oral mucositis at week 12and week 24
Progression-free survival(PFS) | Up to approximately 28 weeks
  The Time from randomization to tumor progression or death due to any cause
Treatment interruption rate | Up to approximately 28 weeks
  Time from the initial administration of TROP2-ADC to treatment interruption

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No